CLINICAL TRIAL: NCT01042834
Title: Impact of Air Pollution on the Autonomic Nervous System Activity and the Presence of Sleep Apnea in Older Subjects: Longitudinal Multicentric Study
Brief Title: Impact of Air Pollution on the Autonomic Nervous System Activity and the Presence of Sleep Apnea in Older Subjects
Acronym: POLLAIR
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Clément CAILLAUX, Centre Hospitalier Universitaire de Saint-Etienne
Other Study IDs: 0508078; DGS 2006/0060 (Other: AFSSAPS)
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2011-01

CONDITIONS: Healthy
Keywords: air pollution; autonomic nervous system; sleep apnea; Heart rate variability; Healthy volunteers
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Air pollution: The subjects will have to live in districts where important atmospheric pollution is established
  Interventions: Other: Air pollution study on healthy volunteers.

INTERVENTIONS:
Other: Air pollution study on healthy volunteers. — The subjects are examined three times:
  * First the volunteers get used to equipments.
  * Second and third the volunteers sleep in a pollution or purified air.
  Other Names: physiopathologic study

SUMMARY:
Impact of air pollution on the autonomic nervous system activity and presence of sleep apnea in older subjects.

DETAILED DESCRIPTION:
The relation between the air pollution and morbidity, cardiovascular mortality was increasing interest. Analyses show an increase of respiratory difficulty, but also cardiac deaths in the daytime when the atmospheric pollution was increased. It was demonstrated that health effects of ambient air pollution in subjects presenting cardiac or lung difficulty were important. Mechanisms show a possible relation to autonomic nervous system (ANS) deactivation and mortality. Particularly, the ageing and ANS reach would be more predictive of cardiovascular events. Thus, we suggest estimating in 60 healthy volunteers from 60 to 80 years old, the impact of the air pollution on the autonomic nervous system activity and sleep apnea consequences.

ELIGIBILITY:
Inclusion Criteria:

* reside in Lyon and Saint-Etienne cities
* security social affiliated or beneficiary
* information note signed

Exclusion Criteria:

* heart rate disorders
* pacemaker
* tabacco addiction or second-hand smoke
* morbid obesity (BMI > 30)
* insulin-dependent diabetes
* chronic disease on treatment
* antiarrythmic treatments

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects will have to live in districts where important atmospheric pollution is established
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Frequency analysis of heart rate variability | inclusion, 1 test night and 2 experimental nights

SECONDARY OUTCOMES:
Analysis of sleep, diurnal somnolence, sleep latency and PRS impact on the life quality. | 1 test night and 2 experimental nights
Hour index quantification of night respiratory events. | 1 test night and 2 experimental nights
Hour index quantification of autonomic awakening during the sleep. | 1 test night and 2 experimental nights

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude BARTHELEMY, MD-PhD, Principal Investigator — CHU de Saint-Etienne
Locations (2):
- France (2):
  - Hospices Civiles de Lyon, Lyon
  - CHU Saint-Etienne, Saint-Etienne